CLINICAL TRIAL: NCT03734562
Title: Randomized Controlled Phase IV Multicentric Trial, Comparing the Efficacy and Safety of Radiofrequency Substrate Ablation of Monomorphic Ventricular Tachycardia vs. Antiarrhyhtmic Drugs in Patients Experiencing Appropriate ICD Shocks
Brief Title: Trial to Evaluate the Efficacy and Safety of Substrate Ablation of Monomorphic Ventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBHGM-0902
Record Dates: First submitted 2017-06-13; First posted 2018-11-08 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Monomorphic Ventricular Tachycardia
Keywords: Ventricular tachycardia; Ischemic cardiomyopathy; Catheter Ablation; Antiarrhythmic drug therapy; ICD
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation; Anti-Arrhythmia Agents; Amiodarone; Sotalol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: ICD therapy analysis and outcome adjudication is performed by physicians blinded to the study group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ablation (Experimental): Substrate-based radiofrequency catheter ablation
  Interventions: Procedure: Ablation
- Antiarrhythmic drug therapy (Active Comparator): Antiarrhythmic drug therapy; amiodarone or sotalol
  Interventions: Drug: Antiarrhythmic drug

INTERVENTIONS:
Procedure: Ablation — Substrate-based radiofrequency catheter ablation
  Other Names: Catheter Ablation
  Arms: Ablation
Drug: Antiarrhythmic drug — Amiodarone or sotalol therapy
  Other Names: Amiodarone, Sotalol
  Arms: Antiarrhythmic drug therapy

SUMMARY:
To compare the efficacy and safety of substrate-based radiofrequency catheter ablation vs. antiarrhythmic drug therapy in patients with ischemic cardiomyopathy and scar-related sustained monomorphic ventricular tachycardia.

DETAILED DESCRIPTION:
Sustained monomorphic ventricular tachycardia remains an important source of morbidity and mortality in patients surviving a myocardial infarction. ICD´s have been proven to reduce mortality in this patients population, nonetheless, recurrent arrhythmia and ICD shocks are known to negatively impact ventricular function and are associated with worsening heart failure and mortality. We devised a controlled, randomized, parallel, single blind, phase IV clinical trial with the aim of comparing the efficacy and safety of substrate-based radiofrequency catheter ablation vs. antiarrhythmic drug therapy in patients with ischemic cardiomyopathy and scar-related sustained monomorphic ventricular tachycardia, implanted with an ICD.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cardiomyopathy, with ischemic myocardial scar
* Sustained monomorphic ventricular tachycardia
* Age > 18 years
* Prior ICD implantation

Exclusion Criteria:

* VT storm
* NYHA functional class IV
* Additional indication for antiarrhythmic drug therapy
* Contraindication for both study drugs (amiodarone and sotalol).
* Uncontrolled myocardial ischemia.
* LV thrombus.
* Non-ischemic VT substrate.
* Contraindications for anticoagulation.
* Prior substrate ablation in the previous 6 months
* Cr > 2.5 mg/dL
* Mitral AND aortic mechanical valvular prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-07; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of death from cardiovascular causes. | 2 years
  - Cause of death will be established by evaluation of medical records by an endpoints adjudication committee. Cardiovascular death includes: sudden death, death due to worsening heart failure or death due to myocardial infarction
Occurrence of appropriate shocks for VT/VF | 2 years
  Occurrence of appropriate shocks for VT/VF VT is measured by ICD interrogation, which is routinely done at the following follow-up visits: after the VT ablation procedure, or in case of suspected arrhythmic symptoms (palpitations, syncope or presyncope).
Occurrence of hospitalization for heart failure | 2 years
  - Hospitalization for heart failure requiring overnight hospital stay and either increased oral diuretics or intravenous diuretics (at least 40 mg od frusemide or 10 mg od torasemide).
Occurrence of severe complication of the ablation procedure. | 2 years
  Occurrence of severe complications of the ablation procedure Will be identified through review of patient clinical reports
Occurrence of interruption of antiarrhythmic drug therapy due to severe side effects | 2 years
  Occurrence of severe complications of the ablation procedure Will be identified through review of patient clinical reports

SECONDARY OUTCOMES:
Number of patients with appropriate ICD therapies | 2 years
  Occurrence of appropriate ICD therapies is measured by ICD interrogation, which is routinely done at the following follow-up visits: after the VT ablation procedure, or in case of suspected arrhythmic symptoms (palpitations, syncope or presyncope). Appropriateness of ICD therapies is established by device-stored electrogram analysis performed by two expert independent electrophysiologists
Number of patients with inappropriate ICD therapies | 2 years
  Occurrence of ICD therapies is measured by ICD interrogation, which is routinely done at the following follow-up visits: after the VT ablation procedure, or in case of suspected arrhythmic symptoms (palpitations, syncope or presyncope).
  Appropriateness of ICD therapies is established by device-stored electrogram analysis performed by two expert independent electrophysiologists
Number of patients with appropriate ICD shocks | 2 years
  Occurrence of ICD shocks is measured by ICD interrogation, which is routinely done at the following follow-up visits: after the VT ablation procedure, or in case of suspected arrhythmic symptoms (palpitations, syncope or presyncope).
  Appropriateness of ICD shocks is established by device-stored electrogram analysis performed by two expert independent electrophysiologists
Number of patients with inappropriate ICD shocks | 2 years
  Occurrence of ICD shocks is measured by ICD interrogation, which is routinely done at the following follow-up visits: after the VT ablation procedure, or in case of suspected arrhythmic symptoms (palpitations, syncope or presyncope).
  Appropriateness of ICD shocks is established by device-stored electrogram analysis performed by two expert independent electrophysiologists
Quality of life measured with the The Short Form (36) Health Survey | 2 years
  Quality of life is measured with the The Short Form (36) Health Survey at pre-specified study follow-up visits (3,6,12,24 months).
  The short-form (36) health survey consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arenal, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General UNiversitario Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Avila P, Berruezo A, Jimenez-Candil J, Tercedor L, Calvo D, Arribas F, Fernandez-Portales J, Merino JL, Hernandez-Madrid A, Fernandez-Aviles F, Arenal A. Bayesian analysis of the Substrate Ablation vs. Antiarrhythmic Drug Therapy for Symptomatic Ventricular Tachycardia trial. Europace. 2023 Jul 4;25(7):euad181. doi: 10.1093/europace/euad181. PMID 37366571
- [Derived] Arenal A, Avila P, Jimenez-Candil J, Tercedor L, Calvo D, Arribas F, Fernandez-Portales J, Merino JL, Hernandez-Madrid A, Fernandez-Aviles FJ, Berruezo A. Substrate Ablation vs Antiarrhythmic Drug Therapy for Symptomatic Ventricular Tachycardia. J Am Coll Cardiol. 2022 Apr 19;79(15):1441-1453. doi: 10.1016/j.jacc.2022.01.050. PMID 35422240